CLINICAL TRIAL: NCT03871738
Title: Efficiency of a Proprioception Work in the Improvement of Sports Performance in Long Jumpers. A Randomized Clinical Trial.
Brief Title: Proprioception in the Improvement of Sports Performance in Long Jumpers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROPIOLJ
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Proprioceptive Disorders
Keywords: Proprioception; Sports performance; Long jump; Physiotherapy; Randomized clinical trial.
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioception training (Experimental): The subjects included in the experimental group will carry out a protocol of proprioception exercises. Each session will last 25 minutes, taking place during 2 sessions a week, in a period of 4 weeks. All interventions will be made before the training session.
  Interventions: Other: Proprioceptive training
- Control (No Intervention): The subjects included in the control group will not receive intervention and will continue to carry out their daily life in the same way as they have done up to now.

INTERVENTIONS:
Other: Proprioceptive training — The intervention to the experimental group will consist of the application of the protocol of proprioception exercises. Before the exercises of the protocol, a warm-up will be carried out that will last 3 minutes and consists of exercises of joint mobility and jumping rope.
  The protocol consists in carrying out two exercises per session, of 10 minutes each. A minute of rest will be implemented between the warm-up and the completion of the protocol, in addition to one minute between the two proprioception exercises in each session. The exercises will vary from week to week, and all the protocol exercises should be done barefoot. The exercise protocol proposed in this study consists of a total of 7 exercises: of unipodal and bipodal support, with unstable surfaces and postural changes.
  Arms: Proprioception training

SUMMARY:
Introduction: In jumping sports the tendinopathies of patellar and Achilles tendon are very frequent. Sports performance is the action that optimizes the relationship between physical abilities and the exercise to be performed. Good proprioceptive work favors the correct execution of the technique in jumping sports.

Aim: To evaluate the effectiveness of the lower limb proprioception exercise in the increase of sports performance, in adults and federated long jumpers Study design: Randomized single-blind multicenter study, with follow-up period. Methods: The 139 subjects included in the study will be randomly assigned to the two study groups: experimental (proprioception protocol) and control (non-intervention group). The intervention will be carried out for 4 weeks, with two weekly sessions, lasting 25 minutes. Three evaluations were carried out (baseline, post-intervention and follow-up). The study variables will be: Proprioception (evaluated by the Romberg test and the SEBT), and sports performance (evaluated with vertical, horizontal jump and competition simulation tests). The analysis of normality will be carried out by the Kolmogorov Smirnof test and in the case of homogeneity of the groups, through the t-student test of related measures and an ANOVA of repeated means, we will calculate the difference between the different evaluations and the effect intra and intersubject.

Expected results. To observe improvement in sports performance, once the proprioceptive exercises have been carried out.

ELIGIBILITY:
Inclusion Criteria:

* Jumping athletes in length
* Female
* With an age range of 18 to 35 years
* Currently participate in regional and / or national competitions.

Exclusion Criteria:

* Not signed the informed consent document
* Practice another sport discipline
* Have some type of medical diagnosis of injury to the lower limb at the time of study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline jump performance of the athlete after intervenion and at month - length of jump | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Using a competition simulator will measure the performance of the athlete, seeking to get as close as possible to the conditions of competition. To carry out this measurement, the athletes will make three full length jumps with approach run of between 14 and 17 steps. Previously, the jumpers will perform their usual warm-up and, between jump and jump, they will have an active rest of 10 minutes. The jump will be measured from the tip of the foot of takeoff, on the board of beaten, to the mark of the sand using a tape measure. The unit of measurement is the centimeter (the greater the distance, the greater the athlete's performance).

SECONDARY OUTCOMES:
Change from baseline jump performance of the athlete after intervenion and at month - vertical jump test | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Through the vertical jump test we will evaluate the jump performance. This measuring instrument has been shown to have high reliability in the measurement of jump performance [ICC = 0.97]. To carry out the evaluation, each subject will perform a practice jump before the test to be measured. The athlete will be placed with both feet resting on the ground, and a shoulder-width apart and a 90º knee flexion, requesting him to make a maximum vertical jump using the arms. The height of the jump will be determined with a tape measure attached to the wall and the chalk mark that the athlete makes in his jump. Each subject will make two jumps and the best score will be chosen for the analysis. The unit of measurement is the centimeter (the greater the distance, the greater the athlete's performance).
Change from baseline jump performance of the athlete after intervenion and at month - horizontal jump test | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Through the horizontal jump test the performance of the athlete will be measured. This measuring instrument has a high intraclass correlation [ICC = 0.93]. The starting position of the athletes will be with both feet resting on the ground, with a shoulder-width apart, following a line marked on the ground. The hands will be placed in neutral position, asking the subjects to make a countermovement with the legs and arms jumping horizontally as much as possible. Finally, they should fall into the sand pit with both feet, registering the horizontal distance between the start line and the heel. The athletes may perform two jumps, being estimated as the value of the evaluation, the best score of both. The unit of measurement is the centimeter (the greater the distance, the greater the athlete's performance).
Change from baseline proprioception after intervenion and at month - unipodal Romberg test | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The unipodal Romberg test is the measuring instrument that will be used for the evaluation of proprioception. It consists of asking the athlete to stand with unipodal support, preferably barefoot and with arms on the sides of the body, maintaining the posture without leaning on their hands. The evaluator, at his side, will be attentive to prevent the athlete from falling due to loss of balance. First you will observe the ability to stay in the position with your eyes open for 5-10 seconds, and if there is postural stability with your eyes open, you will be asked to close your eyes for 20-30 seconds. The unit of measurement of the test is temporary (seconds), indicating a higher score a better proprioception.
Change from baseline proprioception after intervenion and at month - Star Excusion Balance Test | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The Star Excusion Balance Test will be used to evaluate proprioception. This test consists of placing a tape measure on the ground, forming an eight-pointed star, with a 45º separation between them. The patient will be placed with unipodal support in the center of the star, and with the foot in the air you should try to touch as far as possible each line of the star. The evaluator will record the measurement of each line. Each athlete will perform the test three times with each leg, and the evaluator will take the average of those three measurements. The unit of measure is the centimeter, where a greater distance indicates better proprioception.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain